CLINICAL TRIAL: NCT01291134
Title: PureGen Osteoprogenitor Cell Allograft: A Radiographic Analysis of Rate and Quality of Fusion in Patients Undergoing Anterior Cervical Discectomy and Fusion (ACDF)
Brief Title: PureGen: Radiographic Analysis of Fusion for ACDF
Status: Terminated | Type: Observational
Why Stopped: Product is no longer on the market
Sponsor: Alphatec Spine, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO-000053
Record Dates: First submitted 2011-02-04; First posted 2011-02-08 (Estimated); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Cervical Degenerative Disc Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cervical Degenerative Disc Disease: Subjects suffering from symptoms of cervical degenerative disc disease in one to four contiguous levels between C3 and T1.
  Interventions: Biological: PureGen Osteoprogenitor Cell Allograft

INTERVENTIONS:
Biological: PureGen Osteoprogenitor Cell Allograft — PureGen Osteoprogenitor Cell Allograft.

SUMMARY:
The purpose of this study is to evaluate the rate and quality of spinal fusion utilizing PureGen Osteoprogenitor Cell Allograft in Anterior Cervical Discectomy and Fusion (ACDF).

DETAILED DESCRIPTION:
This is a prospective, multi-center, post-market, observational study assessing subjects undergoing cervical interbody fusion surgery to treat cervical degenerative disc disease (DDD)

Patients diagnosed with cervical degenerative disc disease will be screened for enrollment based on inclusion and exclusion criteria outlined in this protocol. Subjects who are successfully screened and sign an informed consent will undergo ACDF surgery utilizing PureGen, Alphagraft ProFuse Demineralized Bone Scaffold (DBS), a radiolucent cervical interbody spacer, and Trestle or Reveal Anterior Cervical Plating System (plate and screw fixation system).

Subjects will be followed at 6- weeks, 3-, 6-, and 12-month post-operative visits. Standard radiographs will be taken at these visits to assess fusion rate and quality. SF-12, NDI and VAS self assessment questionnaires and neurological exams will be administered to measure pain and function scores. A computerized tomography scan will be taken at the 6 month post operative exam to further assess rate and quality of fusion. A conditional 12-month post operative CT may also be taken. Procedure related and device related adverse events will be monitored throughout the study.

Outcome data will be compared to published and/or retrospective data for the standard of care for DDD patients undergoing ACDF.

ELIGIBILITY:
Inclusion Criteria:

* Persistent neck and/or arm pain consistent to symptomatic cervical degenerative disc disease
* Moderate Neck Disability Index
* Unresponsive to conservative treatment for at least 6 weeks

Exclusion Criteria:

* More than 4 levels requiring surgical treatment
* Prior failed fusion surgery at the index level(s)
* Systemic or local infection in the disc or cervical spine, past or present
* Active systemic disease
* Osteoporosis, osteomalacia, or other metabolic bone disease that would significantly inhibit bone healing
* Known or suspected history of alcohol and/or drug abuse
* Involved in pending litigation or worker's compensation relating to the spine
* Pregnant or plans to become pregnant during the duration of the study
* Insulin-dependent diabetes mellitus
* Life expectancy less than study duration
* Any significant psychological disturbance that in the opinion of the Investigator could impair consent process or ability to complete self-assessment questionnaires
* BMI greater than 40
* Undergoing chemotherapy or radiation treatment, or chronic use of oral or injected steroids or prolonged use of non-steroidal anti-inflammatory drugs
* Known history of hypersensitivity or anaphylactic reaction to dimethyl sulfoxide (DMSO).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects suffering from symptoms of cervical degenerative disc disease (DDD) in one to four contiguous levels between C3 and T1.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-02; Primary Completion 2012-02 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Fusion | 12 months
  Proportion of subjects with fusion at the 12-month visit

CONTACTS AND LOCATIONS:
Overall Officials: Bita P. Ghadimi, Study Director — Alphatec Spine, Inc.
Locations (4):
- United States (4):
  - Alphatec Spine Inc., Carlsbad, California
  - Middletown, Connecticut
  - Greensboro, North Carolina
  - Raleigh, North Carolina